CLINICAL TRIAL: NCT01745302
Title: Study of Chinese Medicine Plus EGFR-TKI Versus EGFR-TKI in Advanced Pulmonary Adenocarcinoma: a Randomized Double-blind Controlled Clinical Trial
Brief Title: Efficacy Study of Chinese Medicine Plus EGFR-TKI Versus EGFR-TKI in Advanced Pulmonary Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Ling Xu, Longhua Hospital, Shanghai University of Traditional Chinese Medicine
Other Study IDs: LH126
Record Dates: First submitted 2012-11-22; First posted 2012-12-10 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: lung cancer; traditional Chinese medicine; EGFR-TKI
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TCM plus EGFR-TKIs: TCM:oral granules,YangYinFang or YiQiFang or YiQiYangYinFang,four packages,twice a day, six months; EGFR-TKIs:oral tablet,Gefitinib 250mg daily or Erlotinib 150mg daily or Icotinib 125 mg three times a day ，until progression or unacceptable toxicity;
  Interventions: Drug: TCM; Drug: EGFR-TKI
- Placebo plus EGFR-TKIs: TCM Placebo:oral granules,YangYinFang or YiQiFang or YiQiYangYinFang,four packages,twice a day ,six months; EGFR-TKIs:oral tablet,Gefitinib 250mg daily or Erlotinib 150mg daily or Icotinib 125 mg three times a day until progression or unacceptable toxicity;
  Interventions: Drug: EGFR-TKI

INTERVENTIONS:
Drug: TCM — TCM: In China,TCM herbs are given on the basis of the TCM syndrome differentiation as diagnosed by the TCM herbal specialist. Prescriptions formulated into granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe.The herbal treatment is adapted to the syndromes.
  Other Names: YangYinFang:four packages twice a day; YiQiFang :four packages twice a day; YiQiYangYinFang:four packages twice a day
  Groups: TCM plus EGFR-TKIs
Drug: EGFR-TKI — Erlotinib 150 mg oral once a day or Gefitinib 250 mg oral once a day or Icotinib 125 mg oral three times a day
  Other Names: Erlotinib:150 mg oral, once a day,Tarceva; Gefitinib:250 mg oral, once a day,Iressa; Icotinib:125 mg oral,three times a day,Conmana

SUMMARY:
The investigators performed a randomized, double-blind controlled, prospective study method on observation of Traditional Chinese Medicine combined with targeted therapy to prolong the efficacy of long-term survival of advanced pulmonary Adenocarcinoma patients.The investigators plan to involve 404 cases for observation in 3 years (202 cases for each group), expecting that integrated TCM combined with targeted therapy has a better efficacy on prolonging progression-free survival time, overall survival, improving QOL of patients than that of targeted therapy.

DETAILED DESCRIPTION:
At present, the third generation of platinum-based regimens (NCCN clinical practice guidelines recommended the use of vinorelbine or gemcitabine, or Taxol, etc.) is the first-line treatment for advanced lung cancer patients. Its effective rate is 20-30%, the median survival time is 7-9 months, 1-year and 2-year survival rate is 31-36% and 10-13% respectively. The efficacy has reached the platform and it is difficult to have more breakthroughs. Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) such as Iressa and Erlotinib have proved effective in first or second line therapy for advanced non-small cell lung cancer(NSCLC).First-SIGNAL and IPASS research have laid first-line status for gefitinib in treatment of NSCLC and the progression-free survival time was maintained at 9-10 months. EGFR-TKIs treatment is simple, well tolerated, drug side effects, etc. There are also a rash, diarrhea and other adverse reactions, affecting the quality of life of patients with serious or even give patients a great deal of pain.Literature and our preliminary studies have shown that traditional Chinese medicine (TCM) can prolong survival time and improve quality of life QOL, but high-level evidences are needed.

The investigators perform a randomized, double-blind controlled, prospective study in Advanced Pulmonary Adenocarcinoma patients with stage Ⅲa～Ⅳ. Patients are randomized over observational group (TCM granules plus first-line targeted therapy and TCM granules plus second-line targeted therapy ), and control group (TCM placebo plus first-line targeted therapy and TCM placebo plus second-line targeted therapy). The investigators will observe 6 months and after that regular follow-up will be arranged. The primary efficacy assessments are: PFS (progression-free survival）; Secondary efficacy assessments are: (1) OS(overall survival); (2) Objective response rate; (3) TTP（Time-to-Progression）; (4) QOL (Functional Assessment of Cancertherapy-lung, FACT-L4.0 scales;Lung Cancer Symptom Scale,LCSS); (5)other efficacy assessments are: 1) TCM symptoms changes; 2) Toxicity, side effects and security of the treatments will be assessed at the same time. The investigators expect that integrated TCM combined with targeted therapy has a better efficacy on prolonging progression-free survival time, overall survival, improving QOL of patients than that of targeted therapy. Therefore our study can provide evidences for optimizing and promoting integrated TCM combined with Western Medicine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed of stage IIIa-IV NSCLC with adenocarcinoma histology;
2. Patient with mutated EGFR will subject to first line target thearapy；patients received at least one cycle platinum-containing chemotherapy regimens with disease progression/recurrence， or intolerant/refuse to proceed with chemotherapy will explore second line target therapy;
3. Physical status score (ECOG PS) ≤ 2 scores;
4. Age ≥18 years old;
5. Estimated life expectancy of at least 12 weeks;
6. Participants have no major organ dysfunction: hemoglobin ≥9 g/dL, absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥100 *109/L,bilirubin ≤1.5ULN, alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 upper limited number(ULN) (AP, AST, ALT ≤5ULN is acceptable if liver has tumor involvement).INR≤1.5, APTT in the normal range( 1.2DLN-1.2ULN),creatinine ≤1.5ULN;
7. Informed consent from the patient.

Exclusion Criteria:

1. Patient with other malignant tumor except NSCLC 5 years previous to study entry.
2. Wild type EGFR; already receiving targeted treatment or other anticancer treatment such as palliative radiotherapy if it was not finished over 4 weeks or operation was not over 4 weeks before the first drug administration ;
3. Estimated life expectancy less than 12 weeks;
4. Brain metastasis (controlled brain metastasis and steroid free need is excluded).
5. History of cardiovascular disease: Congestive Heart Failure > grade II in NYHA. Unstable angina patients (have angina symptoms in rest) or a new occurrence of angina (began in the last 3 months) or myocardial infarction happens in the last 6 months;
6. Pregnant or child breast feeding women;
7. Mental or cognitive disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pulmonary adenocarcinoma patients with stage Ⅲa～Ⅳ; TCM syndromes are deficiency of Yin, deficiency of Qi and deficiency of both Qi and Yin.
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 months

SECONDARY OUTCOMES:
Overall response rate(ORR) | 2 months
overall survival(OS) | 2 months
Time-to-Progression(TTP) | 2 months
quality of life(QOL), | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Ling Xu, MD & PhD, Principal Investigator — Longhua Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiao L, Xu J, Sun J, Chen Z, Gong Y, Bi L, Lu Y, Yao J, Zhu W, Hou A, Feng G, Jia Y, Shen W, Li Y, Zhang Z, Chen P, Xu L. Chinese Herbal Medicine Combined With EGFR-TKI in EGFR Mutation-Positive Advanced Pulmonary Adenocarcinoma (CATLA): A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. Front Pharmacol. 2019 Jul 2;10:732. doi: 10.3389/fphar.2019.00732. eCollection 2019. PMID 31333456